CLINICAL TRIAL: NCT01071135
Title: Effects of Quetiapine XR in Schizophrenic Patients With Cannabis Abuse and/or Cannabis Induced Psychosis -Pilot Study-
Brief Title: Quetiapine XR in Schizophrenic Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Planned number of 30 subjects could not be recruited during recruitment phase.
Sponsor: Hannover Medical School (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Wolfgang Dillo, MD, Hannover Medical School
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1443C00018
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Quetiapine XR (Experimental)
  Interventions: Drug: Quetiapine XR

INTERVENTIONS:
Drug: Quetiapine XR — Quetiapine XR (Seroquel Prolong®) extended-release tablets à 50 mg und 200 mg. Seroquel Prolong® should be administered as the only neuroleptics preferably once daily, preferably in the evening. The recommended initial dose is 200 mg/day. Patients should be titrated within a dose range of 400 - 800 mg/day depending on the response and tolerance of the individual patient. Dose increases can be made at intervals as short as 1 day and in increments of up to 200 mg/day. Seroquel Prolong® tablets should be swallowed whole and not split, chewed or crushed.

SUMMARY:
The purpose of the study is to determine the effect of Quetiapine in patients with schizophrenia induced by cannabis abuse.

DETAILED DESCRIPTION:
To evaluate the effect of quetiapine on positive and negative symptoms of schizophrenia on schizophrenic patients associated with cannabis abuse and patients with psychotic disorders through cannabis abuse.

ELIGIBILITY:
Inclusion Criteria:

1. Females and/or males aged 18 to 60 years.
2. Provision of written informed consent. In case of acute psychosis written informed consent has to be obtained from the legal representative of the patient, if applicable or from two independent physicians not involved in the study. When the patient recovers, the written informed consent has to be signed by the patient itself.
3. A diagnosis of schizophrenia (ICD10: F20.0, F20.1, F20.2, F20.4, F20.5) with associated cannabis abuse and/or psychotic disorders (e.g. schizophrenia) through cannabis (ICD 10: F12.5, F12.7).
4. A score of at least 15 on the positive scale of the PANSS.
5. Female patients of childbearing potential must be using a reliable method of contraception (i.e. contraceptive pill, contraceptive coil, sterilization, hysterectomy) and have a negative blood human chorionic gonadotropin (HCG) test at enrollment.
6. Able to understand and comply with the requirements of the study. In case of acute psychosis only those patients are included that are expected to understand the requirements under healthy conditions.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Any ICD10 F-criteria not defined in the inclusion criteria.
3. Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to themselves or others.
4. Known intolerance or lack of response to quetiapine fumarate as judged by the investigator.
5. Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrollment, including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir.
6. Use of any of the following cytochrome P450 3A4 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids.
7. Patients who require treatment with one or more additional neuroleptics to quetiapine.
8. Administration of a depot antipsychotic injection within one dosing interval (for the depot) before randomisation.
9. Substance or alcohol dependence within 4 weeks prior to enrolment, at enrollment and during the study (except for cannabis, caffeine or nicotine dependence), as defined by DSM-IV criteria.
10. Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment.
11. Unstable or inadequately treated medical illness (e.g. congestive heart failure, angina pectoris, hypertension) as judged by the investigator.
12. An absolute neutrophil count (ANC) of ≤ 1.5 x 109 per liter.
13. Involvement in the planning and conduct of the study.
14. Previous enrollment or randomisation of treatment in the present study.
15. A patient with Diabetes Mellitus (DM) fulfilling one of the following criteria:

    * Unstable DM as defined as enrollment glycosylated haemoglobin (HbA1c) >8.5%.
    * Admitted to hospital for treatment of DM or DM related illness in past 12 weeks.
    * Not under physicians care for DM.
    * Physicians responsible for patient´s DM care has not indicated that patient´s DM is controlled. Physician responsible for patient´s DM care has not approved patient´s participation in the study.
    * Has not been on the same dose of oral hypoglycaemic drug(s) and/or diet for the 4 weeks prior to inclusion. For thiazolidinediones (glitazones) this period should be at least 8 weeks.
    * Taking insulin whose daily dose on one occasion in the past 4 weeks has been more than 10% above or below their mean dose in the preceding 4 weeks.

    Note: If a diabetic patient meets one of these criteria, the patient is to be excluded even if the treating physician believes that the patient is stable and can participate in the study.
16. Previous treatment with study medication within the last 4 weeks prior to enrollment into this study.
17. Participation in another drug trial within 4 weeks prior enrollment into this study or current participation in another clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2009-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Reduction in PANSS total score | within 3 months
  The primary variable will be the proportion of patients with a 30% reduction from screening visit to month 3 in PANSS total score.

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Dillo, MD, Principal Investigator — Hannover Medical School
Locations (3):
- Germany (3):
  - Hannover Medical School, Hanover
  - Krankenhaus Lübbecke, Lübbecke
  - Klinikum Wahrendorff, Sehnde